CLINICAL TRIAL: NCT01167192
Title: Effect of Neoadjuvant Platinum-based Chemoradiation Therapy for Locally Advanced Triple Negative Breast Cancer: Clinical Outcome and Correlation to Biological Parameters
Brief Title: Neoadjuvant Platinum-based Chemoradiation Therapy for Locally Advanced Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201310089
Record Dates: First submitted 2010-07-14; First posted 2010-07-22 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin; Carboplatin; Radiotherapy; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation (Experimental): Cisplatin 75 mg/m^2 IV every 21 days for 4 cycles or Carboplatin AUC 6 IV every 21 days for 4 cycles.
  Radiation beginning cycle 2 day 1 daily for 5-6 weeks 45-50 Gy.
  Recommended mastectomy
  Recommended adjuvant chemotherapy
  -doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 for 14 days for 4 cycles followed by paclitaxel 175 mg/m2 for 14 days for 4 cycles)
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Radiation: Radiation therapy; Procedure: Mastectomy (recommended but not mandatory)

INTERVENTIONS:
Drug: Cisplatin
Drug: Carboplatin
Radiation: Radiation therapy
Procedure: Mastectomy (recommended but not mandatory)

SUMMARY:
The purpose of this study is to determine whether platinum-based chemotherapy (either cisplatin or carboplatin), when given with radiation therapy prior to surgery, is effective in improving response to treatment in triple negative breast cancer patients. This treatment is being studied in this type of breast cancer because it does not respond well to commonly used treatments such as tamoxifen or herceptin.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be > or = 18 years of age
* Patient must be female
* Patient must have primary invasive ductal breast adenocarcinoma that either:

  1. is newly diagnosed, without previous systemic treatment OR
  2. has failed to respond to < or = 4 cycles of neoadjuvant anthracycline based therapy as assessed by clinical exam or imaging studies (mammogram, ultrasound or breast MRI).
* Patient's tumor must be classified as clinically stage T2, T3, or T4 with any N (NX, N0, N1, N2, or N3) prior to any neoadjuvant treatment.
* Patient must have an ECOG Performance Status of < or = 1.
* Patient must have adequate organ function defined as:

  1. Renal Function:

     1. CrCl ≥ 60 ml/min for patients receiving cisplatin
     2. CrCl ≥ 30 ml/min for patients receiving carboplatin.
  2. Liver Function:

     1. ALT, AST, ALK Phos < or = 1.5 x upper limit of institutional normal.
     2. Bilirubin < or = 1.5 x upper limit of institutional normal.
  3. Normal left ventricular function (LVEF > 50%) by MUGA or ECHO.
  4. Hematologic:

     1. Absolute Neutrophil Count > or = 1500/mcl
     2. Platelets > or = 100,000/mcl
     3. Hemoglobin > or = 8.0 g/dl
* Patient must be able and willing to sign informed consent document.

Exclusion Criteria:

* Patient must not have evidence of distant metastasis present by CT, bone scan, or PET-CT. If the bone scan or CT scans demonstrate indeterminate lesions, the nature of these lesions should be further clarified by additional testing such as PET or MRI at the discretion of the treating physician.
* Patients having received neoadjuvant anthracycline based therapy must undergo restaging to exclude distant metastases prior to enrollment.
* Patient must not have had any prior malignancies with the exception of curatively treated basal or squamous carcinoma of the skin or history of previous malignancies, treated with at least greater than 5 years disease free survival.
* Patient's tumor must not express the following biomarkers or must have Allred score < 4 for: estrogen receptor, progesterone receptor, and is not Her2/neu amplified.
* Women of child bearing potential may not be currently pregnant or breastfeeding at time of registration and must agree to use adequate contraception.
* Patient must have > or = grade 2 peripheral neuropathy.
* Patient must have a known hearing impairment (hearing loss or severe tinnitus). Hearing test will be performed at the discretion of the treating physician.
* Patient must not have been previously treated with cisplatin or carboplatin for any condition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Aft, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Cleator S, Heller W, Coombes RC. Triple-negative breast cancer: therapeutic options. Lancet Oncol. 2007 Mar;8(3):235-44. doi: 10.1016/S1470-2045(07)70074-8. PMID 17329194
- [Background] Garber, J., Richardson, A., Harris, L., Miron, A., Silver, D., Golshan, M., Ryan, P., Ganesan, S., Wang, Z., Clarke, K., Inglehart, J., and Winer, E. Neoadjuvant cisplatin in triple negative breast cancer. SABCS, 2006.
- [Background] Bollet MA, Sigal-Zafrani B, Gambotti L, Extra JM, Meunier M, Nos C, Dendale R, Campana F, Kirova YM, Dieras V, Fourquet A; Institut Curie Breast Cancer Study Group. Pathological response to preoperative concurrent chemo-radiotherapy for breast cancer: results of a phase II study. Eur J Cancer. 2006 Sep;42(14):2286-95. doi: 10.1016/j.ejca.2006.03.026. Epub 2006 Aug 8. PMID 16893641
- [Background] Formenti SC, Volm M, Skinner KA, Spicer D, Cohen D, Perez E, Bettini AC, Groshen S, Gee C, Florentine B, Press M, Danenberg P, Muggia F. Preoperative twice-weekly paclitaxel with concurrent radiation therapy followed by surgery and postoperative doxorubicin-based chemotherapy in locally advanced breast cancer: a phase I/II trial. J Clin Oncol. 2003 Mar 1;21(5):864-70. doi: 10.1200/JCO.2003.06.132. PMID 12610186
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to enrollment on 02/04/2011 and closed to enrollment on 09/10/2013.
Groups:
- Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation: Cisplatin 75 mg/m^2 IV every 21 days for 4 cycles or Carboplatin AUC 6 IV every 21 days for 4 cycles.
  Radiation beginning cycle 2 day 1 daily for 5-6 weeks 45-50 Gy.
  Recommended mastectomy
  Recommended adjuvant chemotherapy
  -Doxorubicin 60 mg/m^2 and cyclophosphamide 600 mg/m^2 for 14 days for 4 cycles followed by paclitaxel 175 mg/m^2 for 14 days for 4 cycles)
Period: Overall Study
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Started | 10
Completed | 6
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Insurance denial | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 48 [29 to 73]
Gender [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate as Measured by Number of Participants Who Achieved Complete Response (CR) or Partial Response (PR)
Description: * Complete response (CR) = disappearance of all target lesions, disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial response (PR) = at least a 30% decrease in the sum of the longest diameter (LD) of the target lesions taking as reference the baseline sum LD
Time Frame: Prior to surgery (approximately 12-16 weeks from registration)
Population: 1 patient was removed from study due to treatment related toxicity prior to efficacy evaluation and 1 patient expired prior to efficacy evaluation. These two patients are not included in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 6
Participants
  Pathologic complete response | 3
  Partial response | 3

2. Primary Outcome: Relationship Between Tumor Response and Deficiencies in DNA Repair Mechanisms
Time Frame: Prior to surgery (approximately 12-16 weeks from registration)
Population: The physician who was to perform the correlative laboratory work for the study left the university prior to performing the correlative work for this study.
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Disease Progression
Description: Progression = at least a 20% increase in the sum of the longest diameter of the target lesions taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions, appearance of one or more new lesions, unequivocal progression of existing non-target lesions.
Time Frame: Up to 5 years from registration
Population: There are 8 participants not included in this outcome measure and the reasons are as follows: (1) removed from study due to treatment related toxicity prior to surgery, (1) expired prior to surgery, and (6) did not have progressive disease.
Measure: Median (Full Range); unit: months
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 2
months | 6.5 [1.5 to 11.5]

4. Secondary Outcome: Number of Participants With Surgical Complications
Time Frame: 30 days post surgery (approximately 16-20 weeks from registration)
Population: 1 patient was removed from study due to treatment related toxicity prior to surgery and 1 patient expired prior to surgery. These two patients are not included in this outcome measure.
Measure: Number; unit: participant
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 6
participant | 1

5. Secondary Outcome: Determine the Effect of Neoadjuvant Chemoradiation Therapy in Disseminated Cancer Cells in the Bone Marrow
Time Frame: Up to 15 months from registration
Population: as for outcome 2
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival Rate
Time Frame: Median follow-up was 59.9 months
Population: 1 patient was removed from study due to treatment related toxicity prior to surgery and 1 patient expired prior to surgery. These 2 patients are not included in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 8
percentage of participants | 75

7. Secondary Outcome: Medical Toxicities as Measured by Number of Grade 3 or Higher Adverse Events
Time Frame: 30 days post surgery (approximately 16-20 weeks after start of registration)
Measure: Number; unit: adverse event
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 8
adverse event
  Anemia | 1
  Leukocytosis | 1
  Cardiac arrest | 1
  Pulseless electrical activity | 1
  Sinus bradycardia | 1
  Fever | 1
  Wound infection | 1
  Radiation recall reaction (dermatologic) | 1
  Alanine aminotransferase increased | 1
  Creatinine increased | 1
  Lymphocyte count decreased | 4
  Neutrophil count decreased | 1
  Platelet count decreased | 1
  Weight gain | 1
  Hyponatremia | 1
  Back pain | 1
  Cerebrovascular accident | 1
  Acute kidney injury | 1
  Cellulitis | 1
  Hypertension | 1

8. Secondary Outcome: Successful Development of Animal Models of Triple Negative Breast Cancers as Measured by the Ability to Grow the Tumors in Mice.
Time Frame: At the time of IVAD placement and at the time of surgery
Population: Participants did not have sufficient tissue for this outcome measure to be analyzed.
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 0

9. Secondary Outcome: Successful Development of Animal Models for Triple Negative Breast Cancers as Measured by the Ability to Passage the Tumors in Mice
Time Frame: At the time of IVAD placement and at the time of surgery
Population: Participants did not have sufficient tissue for this outcome measure to be analyzed.
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 0

10. Secondary Outcome: Successful Development of Animal Models in Triple Negative Breast Cancers as Measured by the Ability of the Tumors to Metastasize to Other Organs
Time Frame: At the time of IVAD placement and at the time of surgery
Population: Participants did not have sufficient tissue for this outcome measure to be analyzed.
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 0

11. Secondary Outcome: Successful Development of Animal Models of Triple Negative Breast Cancer as Measured by the Genetic Similarity Between the Primary Tumor and the Tumor in Animals
Time Frame: At the time of IVAD placement and at the time of surgery
Population: Participants did not have sufficient tissue for this outcome measure to be analyzed.
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 0

12. Secondary Outcome: Determine the Effect of Neoadjuvant Chemoradiation Therapy in Disseminated Cancer Cells in the Bone Marrow and the Correlation to Tumor Response
Time Frame: Up to 15 months from time of registration
Population: as for outcome 2
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation (N=8)
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Ataxia (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bacteremia (Infections and infestations) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Cerebral-vascular accident (Nervous system disorders) | 1
Chills (General disorders) | 2
Decreased lymphocytes (Investigations) | 2
Decreased platelets (Investigations) | 1
Dysarthia (Nervous system disorders) | 1
Fever (General disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Increased creatinine (Investigations) | 2
Increased international normalized ratio (INR) (Investigations) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pulseless electrical activity (Cardiac disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
Acute renal injury (Renal and urinary disorders) | 1
Alkaline phosphatase increased (Investigations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Cisplatin or Carboplatin AUC 6 & Radiation (N=8)
Alanine aminotransferase increased (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 5
Anxiety (Psychiatric disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Body boils (Skin and subcutaneous tissue disorders) | 1
Body odor (Skin and subcutaneous tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Breast infection (Infections and infestations) | 1
Breast pain (Reproductive system and breast disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Ear clogging (Ear and labyrinth disorders) | 1
Edema - limbs (General disorders) | 3
Edema - trunk (General disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 5
Fever (General disorders) | 1
Headache (Nervous system disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Leg cramping (General disorders) | 1
Lymphedema (Vascular disorders) | 1
Lymphocyte count decreased (Investigations) | 6
Memory impairment (Nervous system disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Neutrophil count decreased (Investigations) | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5
Pharyngitis (Infections and infestations) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Seroma (Injury, poisoning and procedural complications) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Upper respiratory infection (Infections and infestations) | 2
Vomiting (Gastrointestinal disorders) | 2
Watering eyes (Eye disorders) | 1
Weight gain (Investigations) | 1
White blood cell decreased (Investigations) | 4
Wound infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes